## ŚWIADOMA ZGODA RODZICÓW/OPIEKUNÓW PRAWNYCH DZIECKA

biorącego udział w badaniu klinicznym pt.

## "Wpływ pozycji ciała na model defekacji ocenianej przy użyciu manometrii anorektalnej wysokiej rozdzielczości u dzieci"

| Ja niżej podpisany(a) | oświadczam, że |
|---|---|
| przeczytałem/am i zrozumiałem/am powyższe informacje dotyczące opisanego | badania klinicznego |
| oraz otrzymałem/am wyczerpujące, satysfakcjonujące mnie odpowiedzi na zada | ine pytania. Wyrażam |
| dobrowolną zgodę na udział w tym badaniu klinicznym mojego dziecka | a (imię i nazwisko) |
| i jestem świadoma/y faktu, że w każdej chwili mogę wycofać zgodę na udział w | dalszei cześci hadania |
| klinicznego bez podania przyczyny. Przez podpisanie zgody na udział w bad | 2 0 |
| żadnych należnych mi praw. Otrzymam kopie niniejszego formularza opatrzona i | · |

Wyrażam zgodę, by dla kontroli poprawności wykonania badania klinicznego przedstawiciele krajowych, zagranicznych lub międzynarodowych instytucji nadzorujących badanie, mieli wgląd w dane osobowe mojego dziecka oraz dokumentację medyczną (dane dotyczące stanu zdrowia dziecka) pod warunkiem, że są oni związani z badaniem.

Przez podpisanie tego dokumentu potwierdzam również, że zostałem/zostałam poinformowany/poinformowana o sposobie przetwarzania danych z badania i że dane te będą weryfikowane przez ich porównanie z dokumentacją medyczną dziecka oraz że dane te są zbierane jedynie w celu naukowej analizy badania.

Wyrażam zgodę na przetwarzanie danych w tym badaniu zgodnie z obowiązującym w Polsce prawem (Rozporządzenie Parlamentu Europejskiego i Rady (UE) 2016/679 z dnia 27 kwietnia 2016 r. w sprawie ochrony osób fizycznych w związku z przetwarzaniem danych osobowych i w sprawie swobodnego przepływu takich danych oraz uchylenia dyrektywy 95/46/WE). Zgadzam się na przekazanie anonimowych danych mojego dziecka do innych krajów, zarówno w obrębie Europy jak i poza nią.

Dane analizowane przez odnośnie władze, reprezentantów Ministerstwa Zdrowia, agencje rządowe oraz Komisje Bioetyczne dostępne będą jedynie w postaci anonimowej. Zostałem/zostałam poinformowany/poinformowana, iż w przypadku wycofania zgody na udział w badaniu zgromadzone do tej pory dane moga zostać wykorzystane i przetwarzane jako część bazy danych badania.

Zgodnie z art. 13 ogólnego rozporządzenia o ochronie danych osobowych z dnia 27 kwietnia 2016 r.:

- Administratorem Pani/Pana dziecka danych osobowych jest Klinika Gastroenterologii i Żywienia Dzieci Warszawskiego Uniwersytetu Medycznego z siedzibą w Warszawie, ul. Żwirki i Wigury 63A.
- 2. Inspektorem Ochrony Danych w Klinice Gastroenterologii i i Żywienia Dzieci Warszawskiego Uniwersytetu Medycznego jest Marcin Banasiuk, nr tel. 22 317 94 63, adres email marcin.banasiuk@wum.edu.pl. Pani/Pana dziecka dane osobowe przetwarzane będą w celu realizacji badania klinicznego "Wpływ pozycji ciała na model defekacji ocenianej przy użyciu manometrii anorektalnej wysokiej rozdzielczości u dzieci" na podstawie art. 9 ust. 2 lit. a ogólnego rozporzadzenia o ochronie danych osobowych z dnia 27 kwietnia 2016 r.,
- 3. Pani/Pana dziecka dane osobowe mogą być ujawniane wyłącznie:
  - 1) osobom upoważnionym u administratora do przetwarzania danych osobowych,
  - 2) podmiotom przetwarzającym na mocy umowy powierzenia,

- 3) przedstawicielom krajowych, zagranicznych lub międzynarodowych instytucji nadzorujących badanie kliniczne po spełnieniu warunków określonych w Rozdziale V ogólnego rozporządzenia o ochronie danych osobowych z dnia 27 kwietnia 2016 r.,
- 4) innym podmiotom upoważnionym na podstawie przepisów prawa,
- 4. Pani/Pana dziecka dane osobowe przechowywane będą wyłącznie przez okres wymagany przez obowiązujące przepisy prawa,
- 5. posiada Pani/Pan prawo dostępu do treści danych swojego dziecka, prawo do ich sprostowania, usunięcia, ograniczenia przetwarzania, prawo do przenoszenia danych, prawo do wniesienia sprzeciwu i prawo do cofnięcia zgody w dowolnym momencie,
- 6. posiada Pani/Pan prawo wniesienia skargi do Urzędu Ochrony Danych Osobowych, gdy uzasadnione jest, że Pani/Pana dziecka dane osobowe przetwarzane są przez administratora niezgodnie z ogólnym rozporządzeniem o ochronie danych osobowych z dnia 27 kwietnia 2016 r.,
- 7. podanie danych osobowych jest dobrowolne,
- 8. decyzje nie będą podejmowane w sposób zautomatyzowany, nie będzie Pana/Pani dziecko podlegało profilowaniu.

| Rodzic/opiekun prawny: | | |
|---|---|---|
| Imię i nazwisko (drukowanymi literami) | Podpis | Data złożenia podpisu |
| Pacjent >16 rż: | | |
| Imię i nazwisko (drukowanymi literami) | Podpis | Data złożenia podpisu |
| Oświadczam, że omówiłem/omówiłam prze<br>pacjenta/pacjentki używając zrozumiałych,<br>udzieliłem/udzieliłam informacji dotyczący | możliwie prostych sfe | ormułowań oraz |
| Osoba uzyskująca zgodę na badanie | | |
| Imię i nazwisko (drukowanymi literami) | Podpis | Data złożenia podpisu |